CLINICAL TRIAL: NCT00220207
Title: A Randomized Controlled Trial of Diabetes Disease Management Over the Internet
Brief Title: Determining the Effect on Patients of Internet-Based Diabetes Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49154
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Health Education; Information Technology; African Americans; Disease Management; Internet; Patient Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Internet co-management module

SUMMARY:
This grant supports a 12-month randomized controlled trial comparing usual care versus collaborative disease management over the Internet among disadvantaged African-Americans with Type 2 diabetes. The project aims to: (1) determine the effect of case-managed, Web-based diabetes care on glycemic control, health care utilization, self-efficacy, and patient satisfaction; and (2) qualitatively identify enablers of the successful use of computers, the Internet, and e-Health applications by disadvantaged patients.

DETAILED DESCRIPTION:
We propose to conduct a 12-month randomized controlled trial comparing usual care versus chronic disease management over the Internet among disadvantaged African-Americans with type 2 diabetes. Subjects will be recruited from patients receiving primary care at Harborview Medical Center, the County facility administered by the University of Washington in Seattle. As part of a pretest-posttest experimental design, 30 intervention subjects will be trained to use an existing diabetes disease-management module comprising six Web sites that are accessed from home via links displayed within the University's "MyUW" Internet portal. These sites allow patients to:

1. View their entire electronic medical record, the same record used by providers,
2. Upload blood glucose readings stored in a digital meter,
3. Enter medication, nutrition, and exercise information into an online daily diary,
4. Communicate with providers regarding treatment recommendations or other questions using clinical e-mail,
5. Obtain additional information from a traditional patient education site with endorsed content, and
6. Employ a second education site to collaboratively generate action plans intended to enhance self-efficacy.

All data can be viewed by patients and providers in online trended displays that a clinical pharmacist will use to review cases no less often than weekly. As an attention control, 30 subjects will also be trained to use a provided personal computer to access Internet knowledge resources, but will not have access to the case-management services and module being evaluated. By comparing the two groups, we aim to:

1. Determine the effect of case-managed, Web-based diabetes care on glycemic control, healthcare utilization, self-efficacy, and patient satisfaction, and
2. Use semi-structured interviews among a subsample of both trial arms to qualitatively identify enablers of the successful use of computers, the Internet, and e-health applications by disadvantaged patients.

ELIGIBILITY:
Inclusion Criteria:

* African American

Exclusion Criteria:

* non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63
Dates: Start 2003-09; Study Completion 2007-02

PRIMARY OUTCOMES:
Hemoglobin A1c

CONTACTS AND LOCATIONS:
Overall Officials: Harold I. Goldberg, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States